CLINICAL TRIAL: NCT02087176
Title: A Lead-in Phase II Multicentre, Randomised, Double-Blind Study Comparing AZD1775 Plus Docetaxel and Placebo Plus Docetaxel in Previously Treated Non-Small-Cell Lung Cancer Patients
Brief Title: A Placebo Controlled Study Comparing AZD1775+ Docetaxel Versus Placebo+Docetaxel to Treat Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by the sponsor.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6011C00001
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-04

CONDITIONS: Previously Treated Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: interventions — adavosertib; pegfilgrastim; Antimitotic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD 1775, antimitotic, pegfilgrastim (Experimental): AZD 1775, antimitotic agent + pegfilgrastim 21 day Cycle, maximum of 4 cycles
  Interventions: Drug: AZD1775; Drug: Antimitotic Agent; Drug: pegfiligrastim
- Placebo + antimitotic + pegfilgrastim (Placebo Comparator): Placebo + antimitotic+pegfilgrastim 21 day cycle, maximum of 4 cycles
  Interventions: Drug: AZD1775 Placebo; Drug: Antimitotic Agent; Drug: pegfiligrastim

INTERVENTIONS:
Drug: AZD1775 — AZD 1775 + antimitotic agent+ pegfilgrastim, restage every 2 cycles; continue until disease progression or unacceptable toxicity
  Other Names: MK-1775; Neulasta
  Arms: AZD 1775, antimitotic, pegfilgrastim
Drug: AZD1775 Placebo — Placebo (to match dose) + antimitotic+ pegfilgrastim, restage every 2 cycles; continue until disease progression or unacceptable toxicity
  Other Names: MK-1775; Neulasta
  Arms: Placebo + antimitotic + pegfilgrastim
Drug: Antimitotic Agent — The antimitotic is a drug that stops cells from dividing. This leads to cell death. Because cancer cells divide faster than normal cells, they are more likely than normal cells to be affected by this drug.
  Other Names: antiimitotic agent
Drug: pegfiligrastim — Pegfilgrastim is a man-made version of a protein called granulocyte-colony stimulating factor (G-CSF). This protein is made by cells in the body to stimulate the bone marrow to make more infection-fighting white blood cells.Pegfilgrastim is made by attaching filgrastim to a molecule called polyethylene glycol (PEG). This addition helps it stay in the body longer than filgrastim, which means it can be given less often.
  Other Names: Neulasta

SUMMARY:
A Lead-in Phase II Multicentre, Randomised, Double-Blind Study Comparing AZD1775 plus antimitotic agent and Placebo plus an antimitotic agent in Previously Treated Non-Small-Cell Lung Cancer Patients

DETAILED DESCRIPTION:
This multicentre trial consists of an open-labelled single cohort lead-in (Part A) followed by a phase II double-blind, randomised, placebo-controlled comparison of AZD1775 (or placebo) and an antimitotic agent. Review by a central laboratory of fresh tumour or archival tumour samples will be required prior to study entry to assess TP53 mutation status. However, subjects will be allowed to enter the single cohort (Part A) regardless of TP53 mutation status (wild-type or mutant). In addition, patients in the single cohort Part A treatment group will be asked to consent to limited sample collections for assessment of pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria

* Provision of informed consent prior to any study specific procedures
* Histologic or cytologic diagnosis of advanced NSCLC, excluding large cell neuroendocrine, and mixed NSCLC/small-cell histologies
* Failure of one prior platinum-based doublet treatment for advanced NSCLC (either due to progressive disease or toxicity)
* Measurable disease as measured by Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Mandatory availability of tumour tissue (archival or fresh if archival is not available) for TP53 testing
* Male or female ≥18 years-of-age
* Subjects may have received radiation for palliation prior to starting study treatment if they have recovered from the side effects of such therapy
* Absolute neutrophil count (ANC) ≥1500/μL
* Haemoglobin (Hgb) ≥9 g/dL
* Platelets ≥100,000/uL
* Adequate liver function defined as:
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal limits (WNL) or ≤2.5 x upper limit of normal (ULN), if liver metastases are present
* Serum bilirubin WNL
* Adequate renal function
* Ability to swallow oral medication
* Fertile male subjects willing to use at least one medically acceptable form of birth control for the duration of the study and for 2 weeks after treatment stops
* Female subjects who are not of childbearing potential and fertile female subjects of childbearing potential who agree to use adequate contraceptive measures
* Predicted life expectancy ≥12 weeks
* Willingness and ability to comply with study and follow-up procedures
* Ability to understand the investigational nature of this study and give written informed consent
* Most recent chemotherapy ≤21 days or have not recovered from the side effects > Grade 1.
* Use of a study drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of AZD1775
* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting AZD1775 or has not recovered from side effects of such therapy
* Major surgical procedures ≤28 days of beginning AZD1775, or minor surgical procedures ≤7 days
* Known central nervous system (CNS) disease
* Any known hypersensitivity or contraindication to the components of study treatment (AZD1775 and docetaxel)
* Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association [NYHA] ≥ Class 2
* Pregnant or lactating
* Concurrent administration of medications or foods that are strong inhibitors of
* Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the subject to receive protocol treatment
* Presence of other active cancers, or history of treatment for invasive cancer ≤3 years
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Study Chair — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Englewood, Colorado
  - Research Site, Orlando, Florida
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Johnson ML, Dakhil SR, Beck JT, Sadiq A, Menon S, Mugundu GM, Chmielecki J, Spigel DR. Two Phase II Trials of Adavosertib, a Wee1 Inhibitor with Docetaxel or Carboplatin plus Pemetrexed in Non-small-cell Lung Cancer. Target Oncol. 2025 Nov;20(6):967-978. doi: 10.1007/s11523-025-01177-x. Epub 2025 Nov 10. PMID 41212474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 clinical sites in the United States. A total of 32 subjects were enrolled between May 20, 2014 and January 22, 2015.
Pre-assignment Details: 48 participants were screened. 16 did not meet criteria. In Part A, 32 participants were enrolled. The study was terminated early by the sponsor. Part B of the study was not done.
Groups:
- Part A: AZD1775 Plus Docetaxel: Six subject safety lead-in followed by single arm cohort. All patients were to receive AZD 1775 plus Docetaxel in 21 day cycles for a maximum of 4 cycles.
Period: Overall Study
Arm/Group | Part A: AZD1775 Plus Docetaxel
Started | 32
Completed | 0 (The sponsor terminated the study early.)
Not Completed | 32
Not completed — Withdrawal by Subject | 1
Not completed — Death | 10
Not completed — Censored | 19
Not completed — Study Terminated by Sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Part A: AZD1775 Plus Docetaxel
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (9.41)
Age, Continuous [Median (Full Range); unit: Years] | 62.0 [36 to 76]
Age, Customized [Number; unit: Participants]
  < 65 | 18
  >= 65 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: Participants]
  United States | 32
Tobacco Use [Number; unit: Participants]
  Smoker | 29
  Non-Smoker | 1
  Smoking Status Missing | 2
ECOG Performance Status [Number; unit: Participants] — ECOG scores are defined as follows:
  0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1. - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.)
  2. - Symptomatic, < 50% of time in bed during the day.
  3. - Symptomatic, >50% in bed, but not bedbound.
  4. - Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair)
  5. - Death
  Participants
    ECOG Performance Status = 0 | 15
    ECOG Performance Status = 1 | 17

OUTCOME MEASURES:

1. Secondary Outcome: Pharmacokinetic Profile of AZD 1775 in Combination With Docetaxel
Description: Venous blood samples taken for determination of AZD1775, metabolites of 1775 on Cycle 1, Day 1 pre-dose and 2 hours post dose, Cycle 2 Day 1 pre-dose and 2 hours post dose, and Cycle 4 pre-dose and 2 hours post dose. However, the study was terminated early by the sponsor; therefore, pharmacokinetic data were not collected.
Time Frame: Up to projected 20 months, subjects will be restaged after every 2 cycles (every 6 weeks.) continue until disease progression or unacceptable toxicity
Population: The study was terminated early by the sponsor. Pharmacokinetic data have not been analyzed.
Arm/Group | Part A: AZD1775 Plus Docetaxel
Number analyzed (Participants) | 0

2. Primary Outcome: Objective Response Rate
Description: Response evaluation is determined by using Response Evaluation Criteria in Solid Tumours (RECIST v1.1) for target lesions assessed by medical imaging scan (e.g. CT or MRI). The same method of assessment and the same technique was to be used to characterize each identified and reported lesion at baseline and during subsequent imaging procedures. The objective response rate is defined as the percentage of patients with a confirmed best overall response of Complete Response (CR) or Partial Response (PR). Complete Response is defined as disappearance of all target lesions since baseline. Any pathological lymph nodes selected as target lesions must have a reduction in short axis to < 10 mm. Partial Response is defined as at least a 30% decrease in the sum of the diameters of the Target Lesion, taking as reference the baseline sum of diameters.
Time Frame: Up to 20 months
Population: Thirty-two (32) subjects were enrolled in Part A, but the study was terminated early. Patients on-study at the time the study was terminated have been censored.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: AZD1775 Plus Docetaxel
Number analyzed (Participants) | 32
Percentage of Participants | 9.4 [2.6 to 22.5]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event data were collected from the time the first patient received the first dose of investigational drug on May 20, 2014 until the study was closed on May 12, 2015.
Arm/Group | Part A: AZD1775 Plus Docetaxel
Serious Adverse Events (participants affected / at risk) | 17/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: AZD1775 Plus Docetaxel (N=32)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 5
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Leukopenia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) — Grade 4
Abdominal Pain (Gastrointestinal disorders) | 2 (2) — Grade 3
Enterocolitis (Gastrointestinal disorders) | 1 (1) — Grade 3
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 3
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 4
Nausea (Gastrointestinal disorders) | 2 (3) — Grade 3
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3
Asthenia (General disorders) | 2 (2) — Grade 3
Fatigue (General disorders) | 1 (1) — Grade 2
Pneumonia (Infections and infestations) | 1 (1) — Grade 3
Sepsis (Infections and infestations) | 1 (1) — Grade 4
Urinary Tract Infection (Infections and infestations) | 1 (1) — Grade 3
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Failure to Thrive (Metabolism and nutrition disorders) | 1 (1) — Grade 5
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Partial Seizures (Nervous system disorders) | 1 (1) — Grade 1
Syncope (Nervous system disorders) | 1 (1) — Grade 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5
Haemorrhage (Vascular disorders) | 1 (1) — Grade 5
Neutrophil Count Decreased (Investigations) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: AZD1775 Plus Docetaxel (N=32)
Anaemia (Blood and lymphatic system disorders) | 16 (34)
Leukopenia (Blood and lymphatic system disorders) | 7 (8)
Neutropenia (Blood and lymphatic system disorders) | 10 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (24)
Sinus Tachycardia (Cardiac disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 5 (7)
Abdominal Pain, Upper (Gastrointestinal disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 21 (39)
Nausea (Gastrointestinal disorders) | 15 (27)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 14 (19)
Asthenia (General disorders) | 7 (13)
Chest Pain (General disorders) | 2 (2)
Chills (General disorders) | 5 (5)
Face Oedema (General disorders) | 2 (2)
Fatigue (General disorders) | 14 (25)
Malaise (General disorders) | 2 (2)
Mucosal Inflammation (General disorders) | 4 (5)
Oedema Peripheral (General disorders) | 3 (4)
Pain (General disorders) | 7 (10)
Pyrexia (General disorders) | 8 (10)
Pneumonia (Infections and infestations) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (8)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Platelet Count Decreased (Investigations) | 4 (9)
Weight Decreased (Investigations) | 7 (7)
Decreased Appetite (Metabolism and nutrition disorders) | 10 (12)
Dehydration (Metabolism and nutrition disorders) | 10 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Dizziness (Nervous system disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 4 (5)
Neuropathy, Peripheral (Nervous system disorders) | 3 (4)
Syncope (Nervous system disorders) | 2 (2)
Confusional State (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea, Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxsis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Upper Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Hypotension (Vascular disorders) | 6 (7)

LIMITATIONS AND CAVEATS:
The sponsor terminated the study early. The study was closed on May 12, 2015. Part B of the study was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No